CLINICAL TRIAL: NCT04698876
Title: SALUS - Selbsttonometrie Und Datentransfer Bei Glaukompatienten Zur Verbesserung Der Versorgungssituation
Brief Title: Self Tonometry and Transfer of Glaucoma Patients' Data for Improving the Supply Situation
Acronym: SALUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Federal Joint Committee (Other Government); Bielefeld University (Other); Fraunhofer Institute for Applied Information Technology FIT (Unknown); KVWL (Unknown); BARMER (Other); DAK Gesundheit (Other); IKK (Unknown); AOK PLUS (Industry)
Responsible Party: Principal Investigator, Nicole Eter, Chairholder and Head of the Department of Ophthalmology, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01NVF18002
Record Dates: First submitted 2020-11-25; First posted 2021-01-07 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma; Intraocular Pressure; Patient Empowerment; Telemedicine
MeSH Terms: conditions — Glaucoma; Patient Participation | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient measurement of intraocular pressure (Experimental): The intervention group measures its intraocular pressure itself in their home environment for 7 days at 6 a.m., 8 a.m., 12 a.m., 4 p.m., 8 p.m. and 12 p.m. with a self-tonometer (iCareHOME).
  Interventions: Procedure: Self-tonometry by means of ICareHOME; Procedure: Blood pressure
- Stationary measurements of intraocular pressure (Active Comparator): The intraocular pressure of the control group is measured by means of rebound tonometry or Goldmann applanation tonometry in a clinic for minimum 24 hours at 6 a.m., 8 a.m., 12 a.m., 4 p.m., 8 p.m. and 12 p.m.
  Interventions: Procedure: Intraocular measurement by means of rebound tonometry or Goldmann applanation tonometry; Procedure: Blood pressure

INTERVENTIONS:
Procedure: Self-tonometry by means of ICareHOME — Outpatient measurement of intraocular pressure at home
  Arms: Outpatient measurement of intraocular pressure
Procedure: Intraocular measurement by means of rebound tonometry or Goldmann applanation tonometry — Stationary measurement of intraocular pressure in a clinic
  Arms: Stationary measurements of intraocular pressure
Procedure: Blood pressure — Blood pressure measurement for 24 h

SUMMARY:
The SALUS project is developing a new form of care, the application of self-tonometry by the patient itself, and an accompanying electronic case file connecting clinics, doctor's offices and patients.

DETAILED DESCRIPTION:
The SALUS project is developing an outpatient, intersectoral form of care in which patients measure their intraocular pressure in their home environment with a so-called self-tonometer. The measured intraocular pressure values are incorporated into daily pressure profiles, which can be viewed via an electronic case file together with further examination data both by the treating ophthalmologists in the doctor's offices and clinics and by the patients. The new form of care not only supports the telemedical networking of doctors but also increases the compliance by involving the patient in the entire course of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Requirement of a stationary day and night measurement
* Statutory health insurance
* Verified and suspicion of glaucoma diagnosis with suspicion of pressure variations and peaks or not attained target pressure or suspicion of glaucoma progression (H40.1, H40.2 und H42.-)
* Willingness for therapy in one of the participating clinics
* Adequate German language skills
* Signed and dated informed consent for study participation and data transfer
* Legal capacity of the insurant to agree to the study participation

Exclusion Criteria:

* Patients outside the catchment area of the participating clinics
* Covering illnesses in psychiatry, neurology or other indications (e.g. impairment of independence) which make self-tonometry impossible
* Strong communication barriers that do not allow the instruction to carry out the intervention
* Unclear legal capacity of the potential study participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of observed pressure peaks (>30% of the patient-specific target pressure) | 7 days (outpatient) or minimum 24 hours (stationary)
  Measurement of intraocular pressure by means of ICareHOME, rebound tonometry or Goldmann applanation tonometry.

SECONDARY OUTCOMES:
Quality of life (patient-oriented) | Baseline and after 12 months
  By means of a questionnaire, 0: very bad state of health, 1: best possible state of health
Visual field index (VFI) | Baseline and after 9 and 12 months
  By means of perimetry
Mean deviation (MD) | Baseline and after 9 and 12 months
  By means of perimetry
Pattern standard deviation (PSD) | Baseline and after 9 and 12 months
  By means of perimetry
Retinal nerve fiber layer thickness | Baseline and after 12 months
  By means of Optical Coherence Tomography (OCT)/ Heidelberg Retina Tomography (HRT)
Rim volume | Baseline and after 12 months
  By means of Optical Coherence Tomography (OCT)/ Heidelberg Retina Tomography (HRT)
Rim area | Baseline and after 12 months
  By means of Optical Coherence Tomography (OCT)/ Heidelberg Retina Tomography (HRT)
Systolic and diastolic blood pressure | for 24 hours during outpatient and stationary measurements of intraocular pressure
  Long-term blood pressure measurement
Number of inpatient and outpatient health services | 12 month course
  Care provider/ statutory health insurance (SHI) routine data
Costs of health services | 12 month course
  Care provider/ SHI routine data
Number of periods of incapacity for work (unspecific and diagnosis-specific) | 12 month course
  Interview/ SHI routine data
Number of sick pay days | 12 month course
  Interview/ SHI routine data

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Eter, Prof. Dr., Principal Investigator — Chairholder and Head of the Department of Ophthalmology at the University Hospital Muenster
Locations (5):
- Germany (5):
  - Klinikum Dortmund, Dortmund
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Kath. Krankenhaus Hagen, St.-Josefs-Hospital, Hagen
  - Klinikum Luedenscheid, Lüdenscheid
  - University Hospital Muenster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldiges K, Steinmann M, Duevel JA, Gruhn S, Diener R, Leclaire MD, Al-Nawaiseh S, Eter N; SALUS study group. SALUS-a non-inferiority trial to compare self-tonometry in glaucoma patients with regular inpatient intraocular pressure controls: study design and set-up. Graefes Arch Clin Exp Ophthalmol. 2022 Dec;260(12):3945-3955. doi: 10.1007/s00417-022-05759-7. Epub 2022 Jul 22. PMID 35867146
- See also: SALUS Homepage — http://www.salus-glaukom.de